CLINICAL TRIAL: NCT00003577
Title: National Breast Cancer Study of Epirubicin + CMF v Classical CMF Adjuvant Therapy
Brief Title: Combination Chemotherapy With or Without Epirubicin in Treating Women With Stage I or Stage II Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Birmingham (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066644; CRC-TU-NEAT; EU-98041
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2001-02

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CMF regimen; Cyclophosphamide; Epirubicin; Fluorouracil; Methotrexate; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: CMF regimen
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: methotrexate
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether combination chemotherapy plus epirubicin is more effective than combination chemotherapy alone for stage I or stage II breast cancer.

PURPOSE: This randomized phase III trial is studying combination chemotherapy alone to see how well it works compared to combination chemotherapy and epirubicin in treating women with stage I or stage II breast cancer who have undergone surgery to remove the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare disease-free and overall survival of women with early stage breast cancer treated with adjuvant cyclophosphamide, methotrexate, and fluorouracil with or without epirubicin.
* Compare the quality of life in a subgroup of these patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are stratified according to radiotherapy timing (concurrent versus sequential), nodal status (negative versus 1-3 versus at least 4), age (50 and under versus over 50), grade, and tumor size. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive oral cyclophosphamide on days 1-14 and methotrexate IV and fluorouracil IV on days 1 and 8. Treatment repeats every 4 weeks for 6 courses.
* Arm II: Patients receive epirubicin IV on day 1 every 3 weeks for 4 courses followed by cyclophosphamide, methotrexate, and fluorouracil, as in arm I, for 4 courses.

Some patients may receive radiotherapy during or after chemotherapy. Treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed in a subset of patients (N=500) before chemotherapy starts, at 3 months of treatment, at the end of chemotherapy, and at 6, 12, and 18 months after treatment.

Patients are followed annually for 10 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: Approximately 2,000 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histological confirmation of invasive, early stage breast cancer
* Prior complete excision of tumor required (wide local excision or mastectomy)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Not specified

Sex:

* Female

Menopausal status:

* Pre-, peri-, or post-menopausal

Performance status:

* Not specified

Hematopoietic:

* Adequate bone marrow function

Hepatic:

* Adequate hepatic function

Renal:

* Adequate renal function

Other:

* No prior cancer except for basal cell carcinoma or carcinoma in situ
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Concurrent hormone therapy allowed

Radiotherapy:

* No prior radiotherapy
* Concurrent radiotherapy allowed

Surgery:

* See Disease Characteristics
* No more than 6 weeks since prior surgery to the breast

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 1996-03; Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Earl, MBBS, PhD, FRCP, Study Chair — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- University of Cambridge, Cambridge, England, United Kingdom

REFERENCES:
- [Background] Earl H, Hiller L, Dunn JA, et al.: The National Epirubicin Adjuvant Trial (NEAT) and Scottish Cancer Trials Breast Group (SCTBG) br9601 randomized phase III adjuvant early breast cancer trials: the updated definitive joint analysis. [Abstract] J Clin Oncol 25 (Suppl 18): A-534, 11s, 2007.
- [Background] Poole CJ, Earl HM, Hiller L, Dunn JA, Bathers S, Grieve RJ, Spooner DA, Agrawal RK, Fernando IN, Brunt AM, O'Reilly SM, Crawford SM, Rea DW, Simmonds P, Mansi JL, Stanley A, Harvey P, McAdam K, Foster L, Leonard RC, Twelves CJ; NEAT Investigators and the SCTBG. Epirubicin and cyclophosphamide, methotrexate, and fluorouracil as adjuvant therapy for early breast cancer. N Engl J Med. 2006 Nov 2;355(18):1851-62. doi: 10.1056/NEJMoa052084. PMID 17079759
- [Background] Poole CJ, Earl HM, Dunn JA, et al.: NEAT (National Epirubicin Adjuvant Trial) and SCTBG BR9601 (Scottish Cancer Trials Breast Group) phase III adjuvant breast trials show a significant relapse-free and overall survival advantage for sequential ECMF. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-13, 4, 2003.
- [Result] Earl HM, Hiller L, Dunn JA, Bathers S, Harvey P, Stanley A, Grieve RJ, Agrawal RK, Fernando IN, Brunt AM, McAdam K, O'Reilly S, Rea DW, Spooner D, Poole CJ; NEAT Investigators. NEAT: National Epirubicin Adjuvant Trial--toxicity, delivered dose intensity and quality of life. Br J Cancer. 2008 Oct 21;99(8):1226-31. doi: 10.1038/sj.bjc.6604674. Epub 2008 Sep 16. PMID 18797468
- [Derived] Ali HR, Glont SE, Blows FM, Provenzano E, Dawson SJ, Liu B, Hiller L, Dunn J, Poole CJ, Bowden S, Earl HM, Pharoah PD, Caldas C. PD-L1 protein expression in breast cancer is rare, enriched in basal-like tumours and associated with infiltrating lymphocytes. Ann Oncol. 2015 Jul;26(7):1488-93. doi: 10.1093/annonc/mdv192. Epub 2015 Apr 20. PMID 25897014
- [Derived] Ali HR, Provenzano E, Dawson SJ, Blows FM, Liu B, Shah M, Earl HM, Poole CJ, Hiller L, Dunn JA, Bowden SJ, Twelves C, Bartlett JM, Mahmoud SM, Rakha E, Ellis IO, Liu S, Gao D, Nielsen TO, Pharoah PD, Caldas C. Association between CD8+ T-cell infiltration and breast cancer survival in 12,439 patients. Ann Oncol. 2014 Aug;25(8):1536-43. doi: 10.1093/annonc/mdu191. Epub 2014 Jun 9. PMID 24915873